CLINICAL TRIAL: NCT04976179
Title: Intravenous Versus Oral Iron for Iron Deficiency Anaemia in Pregnant Nigerian Women (IVON): an Open Label, Randomized Controlled Trial
Brief Title: Iron Infusion Into a Vein Compared to Iron Tablet Taken by Mouth for Treating Iron Deficiency Anemia in Pregnancy (IVON)
Acronym: IVON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Lagos, Nigeria (Other)
Collaborators: Aminu Kano Teaching Hospital (Other)
Responsible Party: Principal Investigator, Bosede Bukola Afolabi, Professor, University of Lagos, Nigeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACTR202012843695208; ISRCTN63484804 (Registry Identifier: International Standard Randomised Controlled Trial Number); Investment ID INV-017271 (Other Grant/Funding Number: Bill and Melinda Gates Foundation); 2021-002867-23 (EudraCT Number)
Record Dates: First submitted 2021-07-04; First posted 2021-07-26 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: anaemia in pregnancy; iron deficiency; ferric carboxymaltose; ferrous sulphate; intravenous; oral; side effects; effectiveness
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric carboxymaltose; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using Sealed Envelope software and assigned into 2 parallel study arrms as they are recruited. Those in the FCM group will receive Intravenous Ferric Carboxymaltose (Interventional drug) and those in the FS group will receive Oral Ferrous Sulphate (Standard drug).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCM - Intravenous Ferric carboxymaltose (Experimental): Intravenous Ferric Carboxymatlose administered in a single dose of 20mg/Kg to a maximum of 1000mg in 200mls of infusion given over minimum of 15 - 20 minutes at enrollment.
  Interventions: Drug: Ferric carboxymaltose
- FS -Oral Ferrous sulphate (Active Comparator): Oral Ferrous Sulphate (containing 65mg of elemental iron) to be taken as one 200mg tablet 3 times a day until delivery.
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferric carboxymaltose to be given as an intravenous infusion
  Other Names: Ferinject
  Arms: FCM - Intravenous Ferric carboxymaltose
Drug: Ferrous sulfate — Ferrous sulphate tablet to be taken orally
  Other Names: Fesulf
  Arms: FS -Oral Ferrous sulphate

SUMMARY:
Background: Anaemia in pregnancy is a public health burden with high incidence in Africa. Currently high dose oral iron is recommended for treatment of mild to moderate anaemia and blood transfusion for severe anaemia. The high dose oral iron is often poorly tolerated and associated with several side effects. Various parenteral iron preparations are now available for treatment of iron deficiency anaemia (IDA). The earliest of these, iron dextran is not commonly used because of its potential to cause anaphylactic reactions. Newer preparations have been found to be safer and their use for treatment of IDA is currently being evaluated.

Objective: This study sought out to compare the effectiveness of intravenous ferric carboxymaltose (intervention) versus oral ferrous sulphate (control) for treating IDA in pregnancy and to compare the tolerability, safety and the cost-effectiveness of intravenous versus oral iron among pregnant Nigerian women with moderate and severe IDA at 20-32 weeks' gestation.

Methodology: This study will be a hybrid Type 1 effectiveness-implementation design. 1056 eligible and consenting pregnant women with anaemia at 20 - 32 weeks gestation will be recruited. They will be randomized into either of 2 groups. Group A will have intravenous ferric carboxymaltose 20mg/kg to a maximum of 1000mg in 200mls of normal saline infusion over 15 - 20 minutes at enrolment. Group B will have oral ferrous sulphate 200mg (65mg elemental iron) thrice daily from enrolment till delivery. They will be followed up through delivery and until 6 weeks post partum. Their haemoglobin concentration, full blood count, serum ferritin and serum transferrin will be assayed at specific intervals using standard laboratory techniques. Depression will be assessed at each visit using Edinburg Postnatal Depression Scale. Cost effectiveness analysis will also be done at each visit. The primary outcome measure will be incidence of maternal anaemia and rise in haemoglobin level. Secondary outcome measures will include safety and tolerability of trial drugs, severe maternal events, incidence of infant low birth weight and incidence of depression. Statistical analysis will be done using STATA version 16.0 statistical software (STATACorp, Texas, USA).

DETAILED DESCRIPTION:
1.0 INTRODUCTION Anemia in pregnancy (AIP) remains a critical global health problem especially in low- and middle-income countries (LMICs), affecting 46% of pregnant women in Africa and 49% in Asia. AIP is defined as a venous blood hemoglobin concentration of <11 g/dl in a pregnant woman. Iron deficiency anemia (IDA) is the commonest cause of AIP, accounting for 50-75% of AIP. Antenatal maternal anemia has significant implications on both maternal and neonatal outcomes, including maternal mortality from hemorrhage and morbidity from infections, and neonatal low birth weight and prematurity. It has also been associated with an increased risk of depression.

In most LMICs, including Nigeria, routine treatment of IDA in pregnancy is with oral iron preparations, due to fears of serious adverse reactions from parenteral iron, including anaphylaxis, and the belief that oral iron is equally effective. Parenteral, especially intravenous, iron is also more expensive, and it is not clear whether its benefits are worth the cost. In settings like Nigeria, where most people still pay out-of-pocket for healthcare, cost effectiveness is particularly important. However, apart from the side effects caused by oral iron, it also takes longer to correct the anemia, and in cases where patients are unable to absorb iron, oral intake is rendered ineffective. Reservations on use of parenteral iron have been due largely to experience with high molecular weight iron dextran preparations, which had a relatively high incidence of anaphylactic reactions. Fortunately, there are now several safe parenteral iron preparations, such as iron sucrose, iron polymaltose, ferric carboxymaltose (FCM) and iron isomaltoside.

2.0 AIMS AND OBJECTIVES Aims: To determine the comparative effectiveness of intravenous FCM (intervention) versus oral ferrous sulphate (control) for treating iron deficiency anemia in pregnancy and to compare the tolerability, safety, and the cost-effectiveness of intravenous versus oral iron among pregnant Nigerian women with moderate and severe IDA at 20-32 weeks' gestation. It also aims to evaluate the acceptability, feasibility, and fidelity of use of intravenous FCM for treating IDA.

Objectives

1. To determine effect of intravenous FCM on the prevalence of maternal anemia at 36 weeks' gestation and on increase in hemoglobin concentration 4 weeks after administration, compared with oral ferrous sulphate (FS) in pregnant women with IDA.
2. To determine effect of intravenous FCM on incidence of postpartum hemorrhage, sepsis, shock, need for blood transfusion, prevalence of depression and other maternal clinical outcomes, compared with oral FS in pregnant women with IDA.
3. To determine effect of intravenous FCM on the incidence of low infant birthweight, prematurity, stillbirth, and neonatal mortality, and on breastfeeding and immunization, compared with use of oral FS in pregnant women with IDA.
4. To measure implementation outcomes of intravenous FCM including its acceptability, feasibility, and fidelity in the context in which the trial is being carried out.
5. To determine cost-effectiveness of intravenous FCM compared with oral FS in treatment of IDA in pregnancy.

3.0 STUDY DESIGN: This study is a multicenter, parallel, open label, individually randomized controlled trial, with women allocated in a 1:1 ratio in conjunction with a cost-effectiveness analysis.

3.1 Study setting and site selection: The study will be implemented in two most populated states in Nigeria; Kano State in North-West and Lagos State in South-West zone. One tertiary, two secondary and two primary healthcare facilities have been purposively selected from each state, making 10 targeted facilities based on antenatal patient flow, number of deliveries and proximity of all three levels of care to facilitate an effective two-way referral system.

3.2 Sample size calculations: At 5% significance and precision level, 1,056 pregnant women (528 in each study arm) are required to detect a difference in improvement in prevalence of AIP at term by 14%, between control group (70% corrected) and intervention group (84% corrected), as seen in a multi-country international study in Europe, Asia, and Australia (30) at 90% power, adjusting for 15% attrition and protocol violations (31).

3.3 Randomization: At enrolment, eligible participants will be randomized to one of the two treatment groups using a web-based randomization software known as 'Sealed envelope' in a 1:1 ratio in blocks stratified according to center.

3.4 Study intervention: Eligible pregnant women randomized to intervention arm (FCM) will be admitted on a day care basis for treatment initiation and will be given intravenous FCM in a single dose of 20mg/kg up to a maximum of 1000mg in 200 ml 0.9% sodium chloride infusion over a minimum of 15 - 20 minutes. Thereafter, they will be observed for a minimum of 30 minutes before being allowed to go home.

The pregnant women randomized to the control arm (FS) will be given one 200mg tablet of ferrous sulphate containing 65mg of elemental iron, three times daily till 6 weeks post-delivery. The women will be sent daily reminders by text messages, questioned on compliance at each visit and asked to bring in their empty sachets for sighting and pill count.

After delivery, all study participants will be tested for anemia with Hemocue before discharge. Those with hemoglobin concentration less than 11g/dl will be treated as per standard practice i.e., with FS 200mg tds, vitamin C 100mg tds and folic acid 5mg daily.

All study participants in both arms will receive 5mg folic acid daily, vitamin C 100mg tds, and followed from enrollment till delivery and for 6 weeks post-partum. They will be seen 4-weekly till 28 weeks, 2 weekly till 36 weeks and weekly till delivery and then at 2, 4 and 6 weeks postpartum.

3.5 Malaria Treatment and Prevention: Participants will be screened at enrolment for malaria parasitemia with SD BIOLINE Malaria Ag P.f and treated with Artemisinin based combination therapy if positive for malaria parasite. Thereafter, intermittent preventive treatment for malaria will be administered with three doses of three tablets of Sulphadoxine pyrimethamine (500/25) monthly except if patient is allergic to sulphonamides, in which case, patient will be placed on monthly artemisinin-lumefantrine (treatment dose). All pregnant women will also be given long lasting insecticide treated bed nets and counseled on usage.

3.6 Physical examination: Full physical examinations will be performed at baseline, and at each visit. The initial evaluation will also include measurement of patient's weight and blood pressure.

3.7 Laboratory evaluations: These will include:

* Full blood count at enrollment, 4 weeks post enrollment, 36 weeks' gestation, day of delivery and 6 weeks' postpartum.
* Malaria rapid diagnostic test (RDT) with SD BIOLINE Malaria Ag P.f at enrolment and if symptomatic for malaria at any time.
* Hemoglobin concentration with the Hemocue haemoglobinometer at enrolment and every study visit. The first will be used for enrollment.
* Iron profile: This will comprise serum ferritin, serum iron, total iron binding capacity and transferrin saturation at 4 weeks post enrollment, 36 weeks' gestation, day of delivery and 6 weeks postpartum. Only serum ferritin will be done at enrolment.
* Serum phosphate: maternal phosphate level at enrollment, 4 weeks post enrollment, on day of delivery and 6 weeks postpartum; and cord blood phosphate on day of delivery.

All samples aside point of care tests (POCT) will be analyzed at Synlab (an internationally accredited medical laboratory).

3.9 Visit schedules and assessments

* The participants' subsequent clinic visits will be scheduled to hold every 4 weeks till 28 weeks' gestation and every 2 weeks till 36 weeks, then weekly until delivery. Thereafter, they will be seen at 2, 4 and 6 weeks postpartum. Reminders on appointments will be sent by SMS to all participants 24 hours before scheduled visit.
* Women diagnosed as having depression using Edinburg Postnatal Depression Scale (EPDS) will be referred to a psychiatrist for further management.

4.0 DATA ANALYSIS PLAN Data analysis will be by intention-to-treat. Categorical variables will be expressed as frequencies and percentages. For continuous variables, a Shapiro-Wilk test of normality will be performed, and normally distributed data will be presented as means ± SD, while non-normally distributed data will be presented as median and interquartile range (IQR). The risk of occurrence of IUGR, perinatal death and other key outcome variables will be computed and compared in both groups. A multivariate regression analysis will be performed to determine the odds of each of the key outcomes among women who received the intervention with respect to those who did not, after controlling for common confounders. This will be presented as regression coefficients and their 95% confidence intervals. Level of significance will be set at 5%. Post-regression analysis will be performed to determine the goodness-of-fit of the final model. STATA version15.0 (Stata Corp LP, College Station, TX, USA) will be used for statistical analysis.

5.0 MONITORING PLAN - There will also be a Steering committee, Clinical Trial Monitors, and a Data and Safety Monitoring Committee (DSMC).

6.0 ETHICS AND RESEARCH INTEGRITY: This trial has been registered in Pan African Clinical Trials Registry (PACTR202012843695208), International Standard Randomized Controlled Trial Number registry (ISRCTN63484804) and Nigeria Clinical Trial Registry (NCTR, 86233598).

Ethical approvals have been obtained from the National Health Research and Ethics Committee of Nigeria (NHREC), and HREC of both teaching hospitals and health care boards in both states. All study investigators and site coordinators are GCP certified. The research nurses will also be GCP certified.

All participants will sign informed consent form prior to enrolment. Personal data of each participant will be kept strictly confidential and will be stored securely in a central electronic database. Only authorized personnel will have access to the data of all participants collated centrally. The statistician will be granted access to the electronic database during statistical analysis or at any other time the PI might require her to review the data. All research drugs and investigations relating to the research will be offered free.

This research poses minimal or no risk to both mother and baby. Blood specimen collection might cause minimal discomfort in form of pain and care will be taken to minimize this. The intervention drug FCM is known to be safe in pregnancy and is not expected to have significant adverse effects on participants.

All research staff will be adequately trained to monitor, recognize, and manage any significant adverse drug event. In the rare instance of any moderate/severe adverse drug events such as hypophosphatemia and anaphylaxis, trained research staff will effectively resuscitate and transfer care to higher level health facility for adequate care at no cost to the participant.

All participants will receive other routine medication (malaria prophylaxis, tetanus toxoid prophylaxis and folic acid supplementation) as normally prescribed. Malaria prophylaxis, insecticide treated net and folic acid will be provided to the participants all through pregnancy. The participants will enjoy equal rights and quality care all through the duration of the research.

Environmental issues are not applicable to this study. 7.0 DISSEMINATION STRATEGIES The study findings will be presented at conferences (both international and local). Findings will be published in high impact peer reviewed journals. Charts will be created from findings, and these will be used in counselling pregnant women at the various antenatal clinics on complications associated with anemia and preventive measures that may be employed. The researchers will issue press release on study finding.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 15 to 49 years old between 20*- and 32**-weeks' gestational age.
* Baseline (enrollment) laboratory-confirmed moderate or severe anemia (Hb < 10g/dl).

Exclusion Criteria:

* Medically-confirmed significant bleeding, major surgery or received blood transfusion within the last 3 months.
* Severe symptomatic anemia needing urgent correction with blood transfusion.
* Anemia of other cause besides IDA e.g., Sickle cell anemia.
* Clinically-confirmed malabsorption syndrome.
* Hypersensitivity to any form of iron treatment.
* History of any immune related illness e.g., SLE, Rheumatoid arthritis.
* Preexisting maternal depression or other psychiatric illness.
* Severe allergic reactions such as severe asthma.
* History of severe drug allergy.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant females only are eligible to participate in the proposed research.
Enrollment: 1056 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of maternal anemia at 36 weeks' gestation | Measurement taken at 36 weeks gestational age
  To be collected from data source on number of women with hemoglobin concentration less than 10g/dl as determined by hemocue.
Incidence of preterm delivery | Data will be collected following delivery.
  Measured using data source. Preterm delivery is defined as all births after 28 weeks gestational age but before 37 completed weeks of gestation.

SECONDARY OUTCOMES:
Proportion of patients with side effects or intolerance to medication in FCM vs. FS group, including incidence of hypophosphatemia and severe maternal adverse effects at Day 1 and 4 weeks post enrolment, at 36 weeks gestation and 6 weeks post delivery | Assessment to be done on Day 1 and 4 weeks post enrolment, at 36 weeks gestational age and at 6 weeks post delivery
  Measured using information from data source
Proportion of patients with severe maternal events, specifically, haemorrhage, sepsis, shock and the need for blood transfusion measured using data source at delivery | Measured at delivery
  Measured using information from data source
The incidence of low infant birthweight, prematurity, stillbirth and neonatal mortality, proportion of infants being breastfed at 1, 2 and 4 weeks of life, and receiving BCG, oral polio and hepatitis vaccination in same time period | Measurements will be taken at delivery, 1,2 and 4 weeks post delivery
  Measured using data source. Low infant birthweight is defined as <2.5 kg, prematurity is defined as births at <37 weeks' gestation as dated from the last menstrual period or a first trimester ultrasound scan, and neonatal mortality is defined as birth till 28 days of life.
The incidence of depression linked to emotional well-being of mothers using the validated Edinburgh Postnatal Depression Scale measured at enrolment, 36 weeks gestational age and 7 days post delivery | Measurements taken at enrolment, 36 weeks gestational age and 7 days post delivery
  Measurements will de done using the validated Edinburgh Postnatal Depression Scale (EPDS). Maximum score possible on EPDS is 30. Least possible score is 0. A score of 10 and above will be considered positive for depression.
Maternal hemoglobin levels at 4 weeks post-initiation of treatment | Measurement taken at 4 weeks post-initiation of treatment
  Measured in grams per deciliter (g/dl) using hemocue
Prevalence of maternal iron deficiency at 36 weeks' gestation | Measurement taken at 36 weeks gestational age
  To be collected from data source on number of women with iron deficiency defined by serum ferritin level less than 30ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Bosede B Afolabi, DM(Notts), Principal Investigator — College of Medicine, University of Lagos, Idi-araba, Nigeria
Locations (11):
- Nigeria (11):
  - Kabuga Comprehensive Primary Health Centre, Gwarzo, Kano State
  - Kumbotso Comprehensive Health Centre, Kumbotso, Kano State
  - Aminu Kano Teaching Hospital, Tarauni, Kano State
  - Simpson Primary Health Centre, Ebute-Metta, Lagos
  - Lagos University Teaching Hospital, Idi Araba, Lagos
  - Iwaya Primary Health Centre, Iwaya, Lagos
  - Sheikh Jidda General Hospital, Kano
  - Nuhu Bammali Maternity Hospital, Kano
  - Sharada Primary Health Centre, Kano
  - Mother and Child Centre, Amuwo-Odofin, Lagos, Lagos
  - Lagos Island Maternity Hospital, Lagos, Lagos

IPD SHARING:
Plan to Share IPD: Yes
We will store the data and deposit it in 'Open Science Framework', after approval is obtained from the ethics committee. We will also provide metadata along with the data to describe it. No patient identifier will be included in data shared. Potential new users may access our data including the metadata on the 'Open Science Framework'. We will share the data at the time of publication of our first paper. The assigned DOI number, the OSF website details and our approach to data sharing will be included as an appendix to all publications emanating from this research to facilitate accessibility to our data and metadata. We will also share these at any conference presentation both international and local, and also on our study website to facilitate access to it by other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD sharing will commence at the time of first publication or within 6 months of study completion. The duration of IPD sharing will be 2 years, starting tentatively on 1st January 2024 and ending in 31st December 2025.
Access Criteria: The principal investigator will bear overall responsibility for this data and will be responsible for deciding whether to supply research data to a potential new user. The CMUL HREC will provide an independent oversight function.
  2. Data will be made available at the time of publication, at the latest. Depending on the nature of the data itself, data may be made available earlier, either on an individual basis to interested researchers and/or potential new collaborators.
  3. We will ensure that our informed consent forms clearly spell out and seek consent for future data sharing. However, only de-identified data will be shared. I think we will need to clearly spell out the data sharing process.
  4. All external users will sign and be bound by our data sharing agreements and will not be allowed to use the data for reasons other than stated in their application.
  5. IPD sharing will be by open access on Open Science Framework during the period of IPD sharing.

REFERENCES:
- [Background] WHO. The global prevalence of anemia in 2011. Geneva: World Health Organization. 2011 [Available from: https://apps.who.int/iris/bitstream/handle/10665/177094/9789241564960_eng.pdf,accessed?sequence=1.
- [Background] Balarajan Y, Ramakrishnan U, Ozaltin E, Shankar AH, Subramanian SV. Anaemia in low-income and middle-income countries. Lancet. 2011 Dec 17;378(9809):2123-35. doi: 10.1016/S0140-6736(10)62304-5. Epub 2011 Aug 1. PMID 21813172
- [Background] Parks S, Hoffman MK, Goudar SS, Patel A, Saleem S, Ali SA, Goldenberg RL, Hibberd PL, Moore J, Wallace D, McClure EM, Derman RJ. Maternal anaemia and maternal, fetal, and neonatal outcomes in a prospective cohort study in India and Pakistan. BJOG. 2019 May;126(6):737-743. doi: 10.1111/1471-0528.15585. Epub 2019 Jan 24. PMID 30554474
- [Background] Kang SY, Kim HB, Sunwoo S. Association between anemia and maternal depression: A systematic review and meta-analysis. J Psychiatr Res. 2020 Mar;122:88-96. doi: 10.1016/j.jpsychires.2020.01.001. Epub 2020 Jan 8. PMID 31945502
- [Background] Dama M, Van Lieshout RJ, Mattina G, Steiner M. Iron Deficiency and Risk of Maternal Depression in Pregnancy: An Observational Study. J Obstet Gynaecol Can. 2018 Jun;40(6):698-703. doi: 10.1016/j.jogc.2017.09.027. Epub 2018 Jan 4. PMID 29307706
- [Background] WHO. Treatments for iron-deficiency anemia in pregnancy. 2007 [Available from: https://extranet.who.int/rhl/topics/pregnancy-and-childbirth/medical-problems-during-pregnancy/anaemia-during-pregnancy/treatments-iron-deficiency-anaemia-pregnancy
- [Background] Auerbach M, Gafter-Gvili A, Macdougall IC. Intravenous iron: a framework for changing the management of iron deficiency. Lancet Haematol. 2020 Apr;7(4):e342-e350. doi: 10.1016/S2352-3026(19)30264-9. PMID 32220343
- [Background] Radhika AG, Sharma AK, Perumal V, Sinha A, Sriganesh V, Kulshreshtha V, Kriplani A. Parenteral Versus Oral Iron for Treatment of Iron Deficiency Anaemia During Pregnancy and post-partum: A Systematic Review. J Obstet Gynaecol India. 2019 Feb;69(1):13-24. doi: 10.1007/s13224-018-1191-8. Epub 2019 Jan 17. PMID 30814805
- [Background] WHO. Trends in Maternal Mortality: 2000-2017 2019 [Available from: https://apps.who.int/iris/bitstream/handle/10665/327595/9789241516488-eng.pdf?ua=1
- [Background] National Population Commission Nigeria. National Demographic and Health Survey Nigeria 2018 [Available from: https://dhsprogram.com/pubs/pdf/FR359/FR359.pdf
- [Background] Vanderjagt DJ, Brock HS, Melah GS, El-Nafaty AU, Crossey MJ, Glew RH. Nutritional factors associated with anaemia in pregnant women in northern Nigeria. J Health Popul Nutr. 2007 Mar;25(1):75-81. PMID 17615906
- [Background] Bukar M, Audu B, Sadauki H, El-Nafaty AU, Mairiga A. Prevalence of iron deficiency and megaloblastic anemia at booking in a secondary health facility in north eastern Nigeria. Nigerian Medical Journal. 2009;50(2):33-7.
- [Background] Erhabor O, Isaac I, Isah A, Udomah F. Iron Deficiency Anemia among Antenatal Women in Sokoto, Nigeria. British Journal of Medical and Health Sciences. 2013;1(4):47-57.
- [Background] Ajepe AA, Okunade KS, Sekumade AI, Daramola ES, Beke MO, Ijasan O, Olowoselu OF, Afolabi BB. Prevalence and foetomaternal effects of iron deficiency anaemia among pregnant women in Lagos, Nigeria. PLoS One. 2020 Jan 23;15(1):e0227965. doi: 10.1371/journal.pone.0227965. eCollection 2020. PMID 31971986
- [Background] Okafor I, Ibanga I, Asuquo J. Prevalence of Anemia and Iron Deficiency Anemia among Pregnant Women in a Nigerian Rural Community. Sokoto Journal of Medical Laboratory Science. 2018;3(2):52-8.
- [Background] Stevens GA, Finucane MM, De-Regil LM, Paciorek CJ, Flaxman SR, Branca F, Pena-Rosas JP, Bhutta ZA, Ezzati M; Nutrition Impact Model Study Group (Anaemia). Global, regional, and national trends in haemoglobin concentration and prevalence of total and severe anaemia in children and pregnant and non-pregnant women for 1995-2011: a systematic analysis of population-representative data. Lancet Glob Health. 2013 Jul;1(1):e16-25. doi: 10.1016/S2214-109X(13)70001-9. Epub 2013 Jun 25. PMID 25103581
- [Background] Auerbach M. Commentary: Iron deficiency of pregnancy - a new approach involving intravenous iron. Reprod Health. 2018 Jun 22;15(Suppl 1):96. doi: 10.1186/s12978-018-0536-1. PMID 29945649
- [Background] Pena-Rosas JP, De-Regil LM, Garcia-Casal MN, Dowswell T. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2015 Jul 22;2015(7):CD004736. doi: 10.1002/14651858.CD004736.pub5. PMID 26198451
- [Background] Qassim A, Grivell RM, Henry A, Kidson-Gerber G, Shand A, Grzeskowiak LE. Intravenous or oral iron for treating iron deficiency anaemia during pregnancy: systematic review and meta-analysis. Med J Aust. 2019 Oct;211(8):367-373. doi: 10.5694/mja2.50308. Epub 2019 Aug 22. PMID 31441077
- [Background] Chertow GM, Mason PD, Vaage-Nilsen O, Ahlmen J. On the relative safety of parenteral iron formulations. Nephrol Dial Transplant. 2004 Jun;19(6):1571-5. doi: 10.1093/ndt/gfh185. PMID 15150356
- [Background] Pollock RF, Muduma G. A budget impact analysis of parenteral iron treatments for iron deficiency anemia in the UK: reduced resource utilization with iron isomaltoside 1000. Clinicoecon Outcomes Res. 2017 Aug 10;9:475-483. doi: 10.2147/CEOR.S139525. eCollection 2017. PMID 28848355
- [Background] Wolf M, Rubin J, Achebe M, Econs MJ, Peacock M, Imel EA, Thomsen LL, Carpenter TO, Weber T, Brandenburg V, Zoller H. Effects of Iron Isomaltoside vs Ferric Carboxymaltose on Hypophosphatemia in Iron-Deficiency Anemia: Two Randomized Clinical Trials. JAMA. 2020 Feb 4;323(5):432-443. doi: 10.1001/jama.2019.22450. PMID 32016310
- [Background] Consolidated Framework for Implementation Research (CFIR). Interview Guide Tool 2020 [Available from: https://cfirguide.org/guide/app/#/.
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Demographic Statistics Bulletin. Nigeria: National Bureau of Statistics; 2018.
- [Background] Macrotrends. Lagos, Nigeria Metro Area Population 1950-2020 2020 [Available from: https://www.macrotrends.net/cities/22007/lagos/population.
- [Background] Al RA, Unlubilgin E, Kandemir O, Yalvac S, Cakir L, Haberal A. Intravenous versus oral iron for treatment of anemia in pregnancy: a randomized trial. Obstet Gynecol. 2005 Dec;106(6):1335-40. doi: 10.1097/01.AOG.0000185260.82466.b4. PMID 16319260
- [Background] Breymann C, Milman N, Mezzacasa A, Bernard R, Dudenhausen J; FER-ASAP investigators. Ferric carboxymaltose vs. oral iron in the treatment of pregnant women with iron deficiency anemia: an international, open-label, randomized controlled trial (FER-ASAP). J Perinat Med. 2017 May 24;45(4):443-453. doi: 10.1515/jpm-2016-0050. PMID 27278921
- [Background] Bolarinwa OA. Sample size estimation for health and social science researchers: The principles and considerations for different study designs. Niger Postgrad Med J. 2020 Apr-Jun;27(2):67-75. doi: 10.4103/npmj.npmj_19_20. PMID 32295935
- [Background] Kochhar PK, Kaundal A, Ghosh P. Intravenous iron sucrose versus oral iron in treatment of iron deficiency anemia in pregnancy: a randomized clinical trial. J Obstet Gynaecol Res. 2013 Feb;39(2):504-10. doi: 10.1111/j.1447-0756.2012.01982.x. Epub 2012 Aug 26. PMID 22925176
- [Background] Haider BA, Olofin I, Wang M, Spiegelman D, Ezzati M, Fawzi WW; Nutrition Impact Model Study Group (anaemia). Anaemia, prenatal iron use, and risk of adverse pregnancy outcomes: systematic review and meta-analysis. BMJ. 2013 Jun 21;346:f3443. doi: 10.1136/bmj.f3443. PMID 23794316
- [Background] Chandrasekaran N, De Souza LR, Urquia ML, Young B, Mcleod A, Windrim R, Berger H. Is anemia an independent risk factor for postpartum depression in women who have a cesarean section? - A prospective observational study. BMC Pregnancy Childbirth. 2018 Oct 11;18(1):400. doi: 10.1186/s12884-018-2032-6. PMID 30314455
- [Background] Ehlken B, Nathell L, Gohlke A, Bocuk D, Toussi M, Wohlfeil S. Evaluation of the Reported Rates of Severe Hypersensitivity Reactions Associated with Ferric Carboxymaltose and Iron (III) Isomaltoside 1000 in Europe Based on Data from EudraVigilance and VigiBase between 2014 and 2017. Drug Saf. 2019 Mar;42(3):463-471. doi: 10.1007/s40264-018-0769-5. PMID 30535629
- [Background] Ramsey SD, Willke RJ, Glick H, Reed SD, Augustovski F, Jonsson B, Briggs A, Sullivan SD. Cost-effectiveness analysis alongside clinical trials II-An ISPOR Good Research Practices Task Force report. Value Health. 2015 Mar;18(2):161-72. doi: 10.1016/j.jval.2015.02.001. PMID 25773551
- [Background] Common Terminology Criteria for Adverse Events (CTCAE); version 5.0. Published: November 27, 2017. U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES; National Institutes of Health; National Cancer Institute.
- [Derived] Afolabi BB, Babah OA, Adeyemo TA, Balogun M, Banke-Thomas A, Abioye AI, Akinajo OR, Galadanci HS, Quao RA, Adelabu H, Sam-Agudu NA, Adaramoye VO, Abubakar A, Banigbe B, Olorunfemi G, Benova L, Larsson EC, Annerstedt KS, Hanson C, Thornton J; IVON Trial Investigators. Intravenous versus oral iron for anaemia among pregnant women in Nigeria (IVON): an open-label, randomised controlled trial. Lancet Glob Health. 2024 Oct;12(10):e1649-e1659. doi: 10.1016/S2214-109X(24)00239-0. PMID 39304237
- [Derived] Akinajo OR, Babah OA, Banke-Thomas A, Benova L, Sam-Agudu NA, Balogun MR, Adaramoye VO, Galadanci HS, Quao RA, Afolabi BB, Annerstedt KS. Acceptability of IV iron treatment for iron deficiency anaemia in pregnancy in Nigeria: a qualitative study with pregnant women, domestic decision-makers, and health care providers. Reprod Health. 2024 Feb 13;21(1):22. doi: 10.1186/s12978-024-01743-y. PMID 38347614
- [Derived] Afolabi BB, Babah OA, Akinajo OR, Adaramoye VO, Adeyemo TA, Balogun M, Banke-Thomas A, Quao RA, Olorunfemi G, Abioye AI, Galadanci HS, Sam-Agudu NA. Intravenous versus oral iron for iron deficiency anaemia in pregnant Nigerian women (IVON): study protocol for a randomised hybrid effectiveness-implementation trial. Trials. 2022 Sep 8;23(1):763. doi: 10.1186/s13063-022-06690-2. PMID 36076211